CLINICAL TRIAL: NCT04059380
Title: Evaluation of iMmune Function in Post-surgical and AuToimmune HYpoparathyroidism: The EMPATHY Study
Brief Title: Evaluation of iMmune Function in Post-surgical and AuToimmune HYpoparathyroidism (EMPATHY)
Acronym: EMPATHY
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Andrea M. Isidori, Full Professor, University of Roma La Sapienza
Other Study IDs: EMPATHY
Record Dates: First submitted 2019-08-14; First posted 2019-08-16 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Hypoparathyroidism; Hypoparathyroidism Postprocedural; Hypoparathyroidism Due to Impaired Parathormone Secretion
Keywords: parathormone; hypoparathyroidism; parathyroid; hypocalcemia; immunity; immune function; quality of life; sleep disturbances; parathyroid hormone
MeSH Terms: conditions — Hypoparathyroidism; Hypocalcemia; Parasomnias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Hypoparathyroidism: Patients with Post-Surgical or Autoimmune Chronic Hypoparathyroidism requiring daily calcium and calcitriol therapy
- Healthy Controls: Age-, sex- and BMI- matched patients referring to our center for diagnostic procedures not affected by hypoparathyroidism

SUMMARY:
This is an observational pilot study for the evaluation of immune function, infectious diseases, psychometric status and quality of life in patients with hypoparathyroidism compared to healthy controls.

DETAILED DESCRIPTION:
This is an observational pilot study for the evaluation of immune function, infectious diseases, psychometric status and quality of life in patients with hypoparathyroidism compared to healthy controls.

All patients with Hypoparathyroidism will be on established conventional therapy with calcium supplements and calcitriol. According to guidelines, possible confounding factors (i.e. Vitamin D, serum magnesium levels) will be evaluated at screening visit. Age-, sex- and BMI- matched healthy controls will be enrolled.

Patients and controls will undergo a screening visit (V0) and a baseline visit (V1) in the following month.

The primary outcome will be the immune profiling of patients with hypoparathyroidism compared to healthy controls by the quantification of peripheral blood mononuclear cells (PBMC) subpopulations assessed by flow cytometry.

Secondary Outcome Measures will be:

Functional evaluation of PBMC cytokine secretion assessed by flow cytometry

Evaluation of calcium signaling components expression compared to healthy controls

Evaluation of PTHR1 expression in immune cells compared to healthy controls

Evaluation of inflammatory cytokines production compared to healthy controls.

Evaluation of quality of life compared to healthy controls. Quality of life will be measured by Short Form (SF)-36-Item Health Survey total score, SF-36-Item Health Survey physical component summary score and SF-36-Item Health Survey mental component summary score.

Evaluation of infectious diseases frequencies and severity compared to healthy controls. Infectious diseases will be evaluated by an adaptation of Infectious Diseases Questionnaire (GNC).

Psychometric evaluation by self-administered questionnaires: Beck depression Index, Middlesex Hospital Questionnaire.

Sleep disturbances evaluation by The Pittsburgh Sleep Quality Index (PSQI) self reported questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Previously diagnosed (at least 6 months before enrolment) hypoparathyroidism which required daily calcium (≥1000mg/die) and calcitriol therapy;
* Signed informed consent to participate in the study.

Exclusion Criteria:

* Transient hypoparathyroidism;
* History of neoplasms, radiotherapy or chemotherapy in the last 5 years;
* Clinical or laboratory signs of significant respiratory, hepatobiliary, or pancreatic disease;
* Severe infections, surgery, trauma requiring hospitalization within 3 months before enrolment;
* Severe chronic kidney disease (stage 4-5);
* Any active blood or rheumatic disorders in the last 5 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 20 patients with post-surgical or autoimmune hypoparathyroidism and 20 age-, sex- and BMI- matched controls, referring to our center for diagnostic procedures for suspected other endocrinopathies, not affected by hypoparathyroidism
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Peripheral Blood Mononuclear Cells | baseline
  Number of cells (number per mm3) of peripheral blood mononuclear cell subpopulations

SECONDARY OUTCOMES:
Cell-specific Inflammatory Cytokine expression | baseline
  Cell-specific Cytokine expression by flow cytometry - Composite outcome measure of Tumor Necrosis Factor α (TNFα), Transforming Growth Factor-β (TGF-β) and Interferon-γ (IFN-γ) intracellular concentration
PTHR1 expression | baseline
  Measurement of PTHR1 expression by Prime Flow RNA assay
Inflammatory cytokines levels | baseline
  Chemiluminescence measurement of TNFα, TGF-β and IFN-γ serum concentrations.
Infectious diseases frequency and severity | baseline
  Frequencies and severity of infectious diseases will be evaluated by modified Infectious Diseases Questionnaire (GNC).
  This questionnaire includes questions on infectious diseases of upper and lower respiratory tract, gastrointestinal tract, skin and urogenital tract contracted during the previous 12 months. Questions investigate on the number and duration of infections, necessity of antibiotic or antifungal therapy, hospital stay and days of absence from work. Final score represents the frequency of infections. Moreover, some questions investigate possible susceptible or protective factors for infectious diseases: vaccinations, use of corticosteroids, concomitant diseases, previous appendectomy, tonsillectomy, adenoidectomy, splenectomy or thymectomy.
Calcium Signaling evaluation | baseline
  Composite outcome consisting of simultaneous measurement of calcium channels and related proteins: Cav1, Calcium Release Activating Channel, Stromal Interaction Molecule 1 (STIM1), Calcium release-activated calcium modulator 1 (encoded by Orai1 gene), Inositol trisphosphate receptor, Nuclear factor of activated T-cells, Calcineurin and Nuclear Factor Kappa-Light-Chain-Enhancer of Activated B cells (NF-kB) expression evaluated by Prime Polymerase chain reaction
Quality of life: SF-36-Item Health Survey questionnaire | baseline
  Quality of life will be evaluated by the Physical Component score and the Mental Component score of the self-administered questionnaire SF-36-Item Health Survey questionnaire.
  This questionnaire measures eight scales: physical functioning, role physical, bodily pain, general health (physical component) and vitality, social functioning, role emotional, mental health (mental component).
  Interpretation of the score will be the following: at each item of the questionnaire corresponds a percentage value (from 0% to 100%). The average of the single items constitutes the scale total percentage (from 0% to 100%); missing data are not considered during calculation. High score defines a more favorable health state.
Psychometric evaluation | baseline
  Psychometric evaluation will be assessed by the scores of two self-administered questionnaires: Beck depression Index and Middlesex Hospital Questionnaire.
  Beck depression Index is a 21-item measure of depressive symptoms. Each answer is scored on a scale value (from 0 to 3 points). The global score is obtained adding all single scores, with a range of 0-63. Higher score constitutes worse burden of symptoms (0-13: minimal depression, 14-19: mild depression, 20-28: moderate depression, 29-63: severe depression) Middlesex Hospital Questionnaire is a self-rating inventory measuring aspects of six distinct categories of psychoneurosis and affective status. Considering symptoms gravity or frequency each answer is scored on a scale value (from 0 to 2 points). Category scores derive from the addition of the scores of 8 questions. Specific cut off are used to distinguish between normal and pathological behavior (anxiety 5, phobia 5, obsession 7, somatization 5, depression 4 and hysteria 4).
Sleep disturbances | baseline
  Sleep disturbances will be evaluated by The Pittsburgh Sleep Quality Index (PSQI). This questionnaire contains 19 self-related questions which are combined to create 7 component scores with a range of 0-3 points (0:no difficulty, 3: severe difficulty). Global score is the result to the addition of all component scores with a range of 0-21 points (0:no difficulty, 21: severe difficulty).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Experimental Medicine, "Sapienza" University of Rome, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Puliani G, Hasenmajer V, Sciarra F, Barbagallo F, Sbardella E, Pofi R, Gianfrilli D, Romagnoli E, Venneri MA, Isidori AM. Impaired Immune Function in Patients With Chronic Postsurgical Hypoparathyroidism: Results of the EMPATHY Study. J Clin Endocrinol Metab. 2021 Apr 23;106(5):e2215-e2227. doi: 10.1210/clinem/dgab038. PMID 33484559